CLINICAL TRIAL: NCT04739176
Title: Evaluation of the Therapeutic Benefit of Rehabilitation With Computerized Mirror Therapy for Patients Suffering From Motor Neurological Disorder (FND) of the Upper Limb.
Brief Title: Mirror Therapy Rehabilitation for Motor Functional Neurological Disorders.
Acronym: FND-mirror
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_1094
Record Dates: First submitted 2021-01-26; First posted 2021-02-04 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Functional Neurological Symptom Disorder
Keywords: functional neurological disorder; computerized mirror therapy; actimeter; body schema; quality of life; manual dexterity; single case experimental design; rehabilitation
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One-on-one rehabilitation program (Experimental)
  Interventions: Other: One-on-one rehabilitation program including computerized mirror therapy in addition to standard rehabilitation.

INTERVENTIONS:
Other: One-on-one rehabilitation program including computerized mirror therapy in addition to standard rehabilitation. — atients will be admitted to the day hospital 2 days a week for 9 weeks. They will participate in a one-on-one rehabilitation program conducted by a multidisciplinary team including a physiotherapist, psychomotor therapist, occupational therapist and a physical activity monitor. Patients will also participate in 12 computerized mirror therapy sessions (twice a day, 2 days a week, from week 4 to 6 of the program).

SUMMARY:
Motor functional neurological disorders (FND) correspond to motor symptoms that are unexplained by an organic lesion but are due to cerebral dysfunction. Patients with these disorders have high rates of disability and health care utilization, and their quality of life is as impaired as that of patients with an "organic" disease. Accompanying these patients in their often-complex health journey represents a socio-economic and human challenge that demands interdisciplinary collaboration. Rehabilitation is seen as an important part of the therapy for motor FND. However, further research is needed to refine appropriate interventions and to create evidence-based recommendations. In this study, patients suffering from a functional neurological motor disorder of the upper limb will be included in a novel rehabilitation protocol that includes computerized mirror therapy. The study will used a multiple baseline, across subjects, single-case experimental design (SCED). In this type of design, each subject is his own control, with individual parameters being repeatedly measured in the presence and absence of the intervention of interest (computerized mirror therapy). Computerized mirror therapy could restore the coherence between the motor program and its execution. The investigators hypothesize that this process could re-normalize upper-limb motor activity and that this will have a beneficial impact on manual dexterity, quality of life, and mental representation capacities of the upper limb.

The objective of this project is to use the single case experimental design method to investigate the efficacy of rehabilitation with computerized mirror therapy for patients suffering from motor neurological disorders (FND) of the upper limb.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Included in the PULSES program (University Program of Liaison and Care for Somatoform Etiologies),
* Announcement and explanation of the diagnosis already given to the patient,
* Motivated to participate in the project,
* Diagnosed with any type of motor functional neurological disorder : partial or complete deficits and abnormal movements,
* With a lateralized disorder (limited to one hemi-body) involving at least the upper limb,
* Disorder must primarily involve the distal part of the upper-limb (fingers, wrist),
* Admitted to the day hospital at Henry Gabrielle Hospital during the study,
* Given free, informed consent in writing after being informed orally and in writing of how the study will proceed.

Exclusion Criteria:

* Patients with visual disorders such as uncorrected diplopia, blindness or low visual acuity (corrected or uncorrected),
* Pregnant, parturient and breastfeeding women,
* Patients under a legal protection measure such as guardianship or curatorship
* Patients not affiliated to a social security scheme (French Social Security) or beneficiaries of a similar scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Change in upper limb motor activity | Continuous measurements over 24 hours, 7 days a week, during the 9 weeks of study participation
  The actimeter will quantify the level of motor activity of each upper limb, defined by acceleration (number of movements per day that can be described as involving weak, moderate, or intense acceleration) and the number of continuous activities over a 24 hour period. We will compare the activity of the affected hand across the three experimental phases and between the affected and non-affected hands within each phase.
Change in the evaluation of achievement of the patient's rehabilitation objectives using the Goal Attainment Scale (GAS) | Once a week during patient participation (9 weeks)
  The GAS will be established and graded individually with the patient during the first visit, with a maximum of 2 objectives.
  The GAS produces a quantitative index of patient goal attainment that the patient determines at the beginning of the study with the help of a professional. The GAS is assessed weekly using a 5-point scale of -2 and +2. The scale allows each patient to set functional goals by scaling them gradually. The patient's initial level should be set at a score of -2 and the desired level should be set at 0, with +2 representing achievement beyond their initial goal.

SECONDARY OUTCOMES:
Manual dexterity assessment using the Box and Block Test | Once a week during patient participation (9 weeks)
  The Box and Block test is a simple and quick evaluation of global upper limb motricity with well established validity, test-retest reliability and inter-rater reproducibility.
  The patient must use one hand to move as many cubes as possible from one side of the box to the other in 60 seconds. The 60-second test is repeated one time for each hand. The score is the number of blocks moved from one compartment to the other in 60 seconds and a separate score is established for each hand.
Subjective assessment of quality of life using a visual analog scale | Once a week during patient participation (9 weeks)
  The visual analog scale provides a self-report measure of the burden of symptoms and associated disability.
  Using a graduated, non-numerical scale the subject must move a cursor to the place that best represents their current quality of life. The examiner then transcribes the cursor position into a number between 0 and 10.
Subjective assessment of pain using a visual analog scale | Once a week during patient participation (9 weeks)
  The visual analog scale provides a self-report measure of the burden of symptoms and associated disability.
  Using a graduated, non-numerical scale the subject must move a cursor to the place that best represents their current pain intensity. The examiner then transcribes the cursor position into a number between 0 and 10.
Evaluation of the body's mental representation capacities using a laterality judgement task | Once a week during patient participation (9 weeks) for the mental representation of the hand, once every 3 weeks for other body parts
  An implicit motor imagery task involving judging the laterality of body parts will be used to evaluate the evolution of each patient's mental representation capacities via two parameters : the response time and the percentage of correct answers.
  This evaluation will be conducted using a computer program that presents photos of body parts in different postures and orientations. The patient must judge the laterality of each body part (for example: right or left hand, right or left foot).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Henry Gabrielle - Hospices Civils de Lyon, Saint-Genis-Laval, France